CLINICAL TRIAL: NCT04894240
Title: A Phase I Tolerability, Safety, Pharmacokinetics and Preliminary Efficacy Study of Oral Monepantel in Individuals With Motor Neurone Disease
Brief Title: A Study of Monepantel in Individuals With Motor Neurone Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurizon Therapeutics Limited (Industry)
Collaborators: FightMND (Other); Calvary Health Care Bethlehem (Unknown); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MON-2021-001
Record Dates: First submitted 2021-05-05; First posted 2021-05-20 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease | interventions — monepantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Monepantel treatment arm (Experimental): Monepantel tablets will be administered to participants in this arm daily for 28 days. Dose escalation will occur at the end of each 28 day period according to a modified Fibonacci sequence based upon recommendations from the safety management committee
  Interventions: Drug: Monepantel

INTERVENTIONS:
Drug: Monepantel — Monepantel is provided to individuals living with ALS/MND as a white oval tablet to be administered once a day following meals

SUMMARY:
Amyotrophic lateral sclerosis/ Motor Neurone Disease (ALS/MND) is a rare and invariably fatal neurological disease. ALS/MND has a terribly high burden on patients, family and carers, and carries great socioeconomic burden. Current best treatment options are expensive and attempt to control disease progression and manage symptoms while offering no cure. Better treatments are wanting.

Monepantel is a well-known veterinary drug, registered as a livestock wormicide in 39 countries. The industry collaborator, PharmAust Ltd, has found that monepantel shows off-target activity, inhibiting a cellular signaling system controlled by mammalian target of rapamycin (mTOR). This stops cancer growth and reduces protein accumulation in diseased cells. PharmAust has already tested monepantel in humans and pet dogs in Phase I and II anti-cancer clinical trials, respectively, in Australia. Data from these trials show that monepantel treatment associates with an exceptionally high safety profile, mTOR signaling inhibition and anticancer activity.

Abnormal protein accumulation within motor neurons of the brain associates with the cause of ALS/MND. Inhibition of the mTOR signaling pathway slows disease progression in certain preclinical models of ALS/MND and is suggested to provide synergy with the ALS/MND standard-of-care drug, riluzole. An alternative mTOR inhibitor, rapamycin, is currently the subject of an ALS/MND clinical trial in humans investigating control of disease progression. Monepantel has a different structure to rapamycin and an apparently better safety profile.

This Phase I Clinical Trial hypothesis is that monepantel administration to individuals living with ALS/MND will safely reduce disease associated protein accumulation in motor neurons and provide therapeutic benefit. To test this hypothesis, the safety and tolerability of oral monepantel administration and markers of efficacy will be tested in individuals living with ALS/MND in a dose escalating Phase I/II Clinical Trial. To mitigate risk, only patients with sporadic and certain known familial types of ALS will be eligible. To further mitigate risk, the monepantel starting dose will be reduced a calculated five-fold compared to that already used in human cancer patients and already demonstrated to be safe and effective as an mTOR inhibitor. Dependent upon incremental outcomes, three higher doses may then be tested, each for minimally 28 days with a duration at the optimal dose of at least six months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures and treatment
* Familial or sporadic ALS/MND diagnosed as clinically possible, probable, or definite according to Awaji-shima Consensus Recommendations
* Seated slow vital capacity (SVC) ≥ 3L in males and ≥ 2.5L in females at screening
* Not taking riluzole or on a stable dose of riluzole for at least 4 weeks prior to the screening visit. While on study, subjects are not allowed to start taking riluzole during the study
* Patient has a competent caregiver who can support the patient's involvement in the study, including assisting the administration of study drug
* Adequate bone marrow reserve, renal and liver function:

  1. absolute neutrophil count (ANC) ≥1500/µL;
  2. platelet count ≥ 100,000/µL;
  3. hemoglobin ≥ 9 g/dL;
  4. creatinine clearance ≥ 60 mL/min (Cockroft & Gault formula);
  5. alanine aminotransferase ALT, SGPT) and/or aspartate aminotransferase (AST, SGOT)
  6. ≤ 2 x upper limit of normal (ULN);
  7. total bilirubin ≤ 1.5 x ULN;
  8. serum albumin ≥ 2.8 g/dL
* Women and men with partners of childbearing potential must use effective contraception while on study treatment and women of childbearing potential must have a negative pregnancy test at screening

Exclusion Criteria:

* Inability to swallow oral medications or presence of a gastrointestinal disorder (e.g., malabsorption) deemed to jeopardize intestinal absorption of study drug
* Dependence on mechanical ventilation (invasive or non-invasive, including Continuous Positive Airway Pressure (CPAP) or Bi-level Positive Airway Pressure (BiPAP) for any part of day or night prior to the screening visit. Dependence on mechanical ventilation is defined as being unable to lie flat (supine) without it, unable to sleep without it, or daytime use
* Exposure to any other investigational agent within 3 months prior to the screening visit
* Active gastrointestinal disease within 30 days of the screening visit. Gastro-esophageal reflux disease (GERD) is not considered active gastrointestinal disease and is not exclusionary
* Known immune compromising illness or treatment
* Presence of any of the following clinical conditions:

  1. drug abuse or alcoholism;
  2. unstable cardiac, pulmonary, renal, hepatic, endocrine, or hematologic disease;
  3. active infectious disease;
  4. AIDS or AIDS-related complex;
  5. diagnosis of malignancy within 2 years of screening (adequately treated basal cell or squamous cell carcinoma of skin or non-invasive bladder cancer or carcinoma in situ of the bladder, breast or cervix are allowed;
  6. unstable psychiatric illness defined as psychosis or untreated major depression within 90 days of the screening visit;
  7. neuromuscular disease other than ALS/MND
* Dementia that may affect either outcome measures or patient understanding and/or compliance with study requirements and procedures
* Women and men of childbearing potential not using effective contraception while on study treatment
* Women who are breast-feeding
* Patients at risk of or known to carry a SOD1 mutation or VCP mutation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Determination of Phase 2 Dose | At least 4 weeks
  A recommended phase 2 dose will be determined by the number of participants at each dose level recording dose limiting toxicities
Blood Plasma Pharmacokinetics of Monepantel | 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours and 2, 8, 15, 22 and 29 days after dosing
  Characterise monepantel blood plasma levels following administration to individuals living with ALS/MND
Blood Plasma Pharmacokinetics of Monepantel Sulfone | 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours and 2, 8, 15, 22 and 29 days after dosing
  Characterise monepantel's major metabolite monepantel sulfone blood plasma levels following administration of monepantel to individuals living with ALS/MND

SECONDARY OUTCOMES:
Treatment related changes in peripheral blood mononuclear cell phosphorylated ribosomal protein S6 kinase B1 (RPS6KB1) levels (pharmacodynamics) | From admission to discharge, up to 6 months
  Changes RPS6KB1 phosphorylation levels will assist in determining if the proposed targeted mammalian target of rapamycin (mTOR) pathway is being correctly affected (photostimulated luminescence units)
Treatment related changes in peripheral blood mononuclear cell phosphorylated eukaryotic initiation factor 4 E binding protein 1 (EIF4EBP1) levels (pharmacodynamics) | From admission to discharge, up to 6 months
  Changes EIF4EBP1 phosphorylation levels will assist in determining if the proposed targeted mammalian target of rapamycin (mTOR) pathway is being correctly affected (photostimulated luminescence units)
Treatment-related changes from Baseline on the ALS Functional Rating Scale (ALSFRS) at Week 4 | From admission to discharge, up to 6 months
  The ALS Functional Rating Scale (ALSFRS) is a validated rating instrument for monitoring the progression of disability in patients with amyotrophic lateral sclerosis (ALS). Measurements include: (1) speech (2) salivation (3) swallowing (4) handwriting (5) cutting food and handling utensils (with or without gastrostomy) (6) dressing and hygiene (7) turning in bed and adjusting bed clothes (8) walking (9) climbing stairs and (10) breathing. Possible scores range from 0 (normal function) to 4 (severe loss of function). Change = (Week 4 score - Baseline score)
Treatment-related changes from Baseline in Edinburgh Cognitive and Behavioural Amyotrophic Lateral Sclerosis Screen (ECAS) at Week 4 | From admission to discharge, up to 6 months
  The ECAS-cognitive screen is a validated screen comprises 16 items organized into two sub-scales. An ALS-specific sub-scale taps into the cognitive domains of language, verbal fluency, and executive and social functions. A non-ALS-specific sub-scale specifically assesses memory and visuospatial function. The sub-scales of the ECAS-cognitive screen range, respectively, from 0 to 100 and from 0 to 36. Low scores indicate a greater deficit. Change = (Week 4 score - Baseline score)
Treatment-related changes from Baseline in slow vital capacity (SVC) | From admission to discharge, up to 6 months
  A decline in SVC would indicate a decline in respiratory function and is an important indicator of any clinical progression (L/s)
Treatment-related changes in urinary p75 levels | From admission to discharge, up to 6 months
  Urinary p75 level reflect nerve damage and therefore increased levels would act as a proxy to disease progression (ng/mg creatinine)
Treatment-related changes in 3 Tesla magnetic resonance imaging (MRI) | From admission to discharge, up to 6 months
  MRI is a method used to investigate and exclude conditions that may mimic motor neuron dysfunction (Tesla)
Treatment-related changes in serum neurofilament light (NfL) chain levels | From admission to discharge, up to 6 months
  Serum NfL chain levels correlate with disease progression, so stable NfL levels would correlate with stable disease (pg/ml)
Treatment-related changes in central spinal fluid (CSF) NfL chain levels | From admission to discharge, up to 6 months
  CSF NfL chain levels correlate with disease progression. Levels in individuals living with MND are 5 to 10 fold higher than those of healthy individuals (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mathers, MB ChB, MRCP(UK), FRACP, Principal Investigator — Calvary Health Care Bethlehem; Dominic Rowe, PhD, FRACP, AM, Principal Investigator — Macquarie University, Sydney
Locations (2):
- Australia (2):
  - Macquarie University, Sydney, New South Wales
  - Calvary Health Care Bethlehem, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mislang A, Mollard R, Tapia Rico G, Fairlie WD, Lee EF, Harris TJ, Aston R, Brown MP. A preliminary assessment of oral monepantel's tolerability and pharmacokinetics in individuals with treatment-refractory solid tumors. Cancer Chemother Pharmacol. 2020 Nov;86(5):589-594. doi: 10.1007/s00280-020-04146-5. Epub 2020 Sep 22. PMID 32960289